CLINICAL TRIAL: NCT04389658
Title: Retrospective Observational Study to Determine COVID-19 Contagious and Immunological Status in Asymptomatic Population of Highly Affected Areas
Brief Title: Contagiousness and Immunogenicity Status of COVID-19 in Asymptomatic Population (COVID-19 CONDITION)
Acronym: CONDITION
Status: Completed | Type: Observational
Sponsor: Igenomix (Industry)
Responsible Party: Sponsor
Other Study IDs: IGX1-COV-XS-20-01
Record Dates: First submitted 2020-05-14; First posted 2020-05-15 (Actual); Last update posted 2020-10-09 (Actual); Status verified 2020-10

CONDITIONS: COVID-19
Keywords: SARS-CoV-2; Severe acute respiratory syndrome coronavirus 2; COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Asymptomatic population: Subjects who underwent PCR and ELISA tests for the diagnosis of COVID-19: mainly asymptomatic individuals from three main areas of Spain (Madrid, Barcelona and Valencia) with high impact of COVID-19 that have performed the PCR and ELISA test for the diagnosis of COVID-19 before initiating the work immediately after Spanish lockdown.

SUMMARY:
In late December 2019, a new coronavirus strain emerged in China causing coronavirus disease 2019 (COVID-19). Since then, COVID-19 has become a global pandemic outbreak being declared a "public health emergency of international concern" by the International Health Regulations Emergency Committee of the WHO on January 30, 2020. Several emergency measures have been implemented in different countries such as lockdown, social distancing and testing. However, due to the lack of tests worldwide the real number of affected and/or immunized people remains largely unknown. In this moment, when reopening phases are being undertaken in the majority of countries, the decision to enact any of these measures rests with the judgement of each health care system. However, every country or individual community circumstances may be unique and require contextual consideration based on the severity and time of the pandemic as well as the number of resources available. The present study aims to retrospectively describe the immune and infective spectrum of illness from Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) infection in the general asymptomatic population in three main areas of Spain (Madrid, Barcelona and Valencia) with high impact of COVID-19, right after the lockdown period.

DETAILED DESCRIPTION:
In late December 2019, a new coronavirus strain emerged in Chinese megacity Wuhan. The World Health Organization (WHO) named it Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV2) leading to coronavirus disease 2019 (COVID-19). On January 30, 2020 the International Health Regulations Emergency Committee of the WHO declared the outbreak a "public health emergency of international concern". On March 11, 2020 WHO characterized COVID-19 as a pandemic and on March 14th, the Spanish President COVID-19 outbreak a "national emergency" for second time in 40 years.

In order to fight this unanticipated pandemic, emergency measures have been implemented in different countries such as lockdown, social distancing and testing. Massive community testing to detect early or asymptomatic infections as well as social distancing has been used in certain countries (South Korea, Iceland, etc..) with relatively success. In this sense, Polymerase Chain Reaction (PCR) is considered to be the gold standard to diagnose the infection with SARS-CoV2. On the other hand, Enzyme Linked ImmunoAssay (ELISA) has also been widely used to determine the presence of antibodies (Immunoglobulins M, A and G) and, hence immunological status. Some studies have reported the presence of IgM and IgA antibodies within the first 5 days of clinical symptom onset, while IgG is usually detected on 14 days after symptom onset, with a positive rate of 85.4%, 92.7% and 77.9%, respectively. Moreover, a recent report of reveals that positive detection rate is significantly increased when combined IgM/IgA ELISA assay with PCR for each patient compare with a single quantitative PCR test. In this sense Igenomix has recently obtained the authorisation by the Valencia Community Authority to provide these services after completing the requested process of verification.

In this moment, when reopening phases are planning or even undertaken in the majority of countries, the decision to enact any of these measures rests with the judgement of each health care system. However, every country or individual community circumstances may be unique and require contextual consideration based on three main factors: the severity of the pandemic spread, the measures and timing implemented during the pandemic, and the moment of the post pandemic that this population is in. Therefore, international metrics are urged to guide the re-opening of the post pandemic era in different parts of the world to provide a logical approach to mitigate risk to new outbreaks.

This is a retrospective, observational study in which anonymized data from subjects who already performed PCR and ELISA test for COVID-19 detection at Igenomix, will be used to assess the rate of immunized population as well as the rate of asymptomatic contagious population in three hot spots of Spain (Madrid, Barcelona and Valencia) immediately after the lockdown period. After data collection and processing, once the full anonymization process has been completed, the pool of data will be analyzed with the aim of retrospectively describe the immune and infective spectrum of illness from SARS-CoV-2 infection in the general asymptomatic population in three main areas of Spain (Madrid, Barcelona and Valencia) with high impact of COVID-19. Moreover, other additional descriptive variables such as age, gender, etc will be assessed.

Being an observational retrospective study, the sample size would consist of the complete database of individuals analyzed by ELISA and PCR from areas of Madrid, Barcelona and Valencia representing approximately 1,000 cases. Waiver of informed consent form has been duly authorized by the Ethic Committee in agreement to the local legislation.

No intervention involving patients or their biological material will be required.

ELIGIBILITY:
Inclusion Criteria:

* Mainly asymptomatic individuals from different corporations of urban areas of Barcelona, Madrid and Valencia that have performed the test before initiating the work immediately after Spanish lockdown from the end of April until beginning of May.

Exclusion Criteria:

* There is not exclusion criteria for this study.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Anonymized data produced by Igenomix from previous PCR and ELISA tests of mainly asymptomatic individuals will be used in this study. Approximately, 1,000 cases will be assessed.
Sampling Method: Non-Probability Sample
Enrollment: 1526 (Actual)
Dates: Start 2020-05-07 (Actual); Primary Completion 2020-06-10 (Actual); Study Completion 2020-08-25 (Actual)

PRIMARY OUTCOMES:
Prevalence of contagiousness in asymptomatic individuals by PCR | 2 months
  This outcome measure statistically quantifies the Prevalence of contagiousness in asymptomatic individuals based on the gold standard test (PCR).
  These results will be analysed in order to focus on the best combination to detect the presence of the disease and the immunological stage in this population at the three main areas of Spain (Madrid, Barcelona and Valencia) with high impact of COVID-19.
Ratio of asymptomatic immunized (IgA/IgM and IgG) population | 2 months
  This outcome measure statistically quantifies the rate of immunized (IgA/IgM and IgG) individuals based on the ELISA test.
  These results will be analysed in order to focus on the best combination to detect the presence of the disease and the immunological stage in this population at the three main areas of Spain (Madrid, Barcelona and Valencia) with high impact of COVID-19.

SECONDARY OUTCOMES:
Description of demographic characteristics | 2 months
  Age, gender and location distribution of affected contagious individuals at the three main areas of Spain (Madrid, Barcelona and Valencia) with high impact of COVID-19.

CONTACTS AND LOCATIONS:
Overall Officials: Xavier Santamaria, MD,PhD, Principal Investigator — Igenomix; Carlos Simon, MD,PhD, Principal Investigator — Igenomix
Locations (1):
- Igenomix, Paterna, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No